CLINICAL TRIAL: NCT06404762
Title: Comparison of Subepithelial Connective Tissue Grafts Harvested from the Maxillary Tuberosity or Lateral Palate in the Treatment of Single Maxillary Recession-type Defects
Brief Title: Tuberosity Versus Palatal Connective Tissue Graft on the Treatment of Single Maxillary Recession-type Defects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sıla Çağrı İşler, Assoc Prof, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-21071282-050.99-519910
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-05

CONDITIONS: Gingival Recession, Localized
Keywords: Maxillary Tuberosity; Connective Tissue Graft; Coronally Advanced Flap
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- tSCTG+ CAF (Active Comparator): Single, isolated gingival recessions; excluding molars; at maxilla will be treated with subepithelial connective tissue graft harvested from the maxillary tuberosity in conjunction with a coronally advanced flap
  Interventions: Procedure: tSCTG+ CAF
- pSCTG+ CAF (Active Comparator): Single, isolated gingival recessions; excluding molars; at maxilla will be treated with subepithelial connective tissue graft harvested from the lateral palate in conjunction with a coronally advanced flap
  Interventions: Procedure: pSCTG+ CAF

INTERVENTIONS:
Procedure: tSCTG+ CAF — In the tSCTG group, at the distal end of a second maxillary molar, an incision will be made using a double-bladed scalpel (SKU 10-130-05D; Hu-Friedy, Chicago, IL, USA) bucco-palatally, forming a 1,5 mm thick parallel line. Secondary incisions will be made to separate the graft using a 15c blade on the buccal and palatal sides. Later, the graft will be de-epithelialized extra-orally using a blade
  Arms: tSCTG+ CAF
Procedure: pSCTG+ CAF — In pSCTG group; the graft will be harvested through a single-incision approach at the lateral palatal mucosa
  Arms: pSCTG+ CAF

SUMMARY:
The goal of this randomized clinical study is to assess the root coverage outcomes and patient morbidity following the treatment of single maxillary recession-type defects using a coronally advanced flap (CAF) combined with a subepithelial connective tissue graft (SCTG) harvested from the maxillary tuberosity (MT) versus lateral palate (LP). The secondary objective is to evaluate the histological characteristics of graft compositions harvested from the different regions (MT versus LP).

Therefore, the following questions related to the study are raised:

* Do SCTGs harvested from MT (tSCTG) and LP (pSCTG) exhibit similar root coverage outcomes in the treatment of single maxillary recession-type defects using CAF?
* What are the histological characteristics of tSCTG and pSCTG?

A total of 30 patients who have been referred to the Gazi University Department of Periodontology will be randomly assigned to receive tSCTG or pSCTG in combination with CAF. Clinical measurements will be recorded at baseline, 1, 3, 6, and 12 months after surgeries. Immediately after interventions; a questionnaire evaluating post-operative pain, discomfort, sensitivity, and bleeding will be given to the patients. The amount of non-steroid anti-inflammatory drugs used will be recorded at 1, 2, 3, 7, 14 and 28 days after surgery. Descriptive morphologic analysis of the grafts will be assessed in terms of the presence of inflammatory cells, connective tissue cellularity, vascularization, adipose tissue, and collagen structure.

DETAILED DESCRIPTION:
The treatment of gingival recessions using the coronally advanced flap (CAF) in combination with palatal subepithelial connective tissue graft (pSCTG) is highly predictable and frequently accepted in periodontal plastic-aesthetic surgeries. However, due to its limitations and disadvantages, clinicians often use grafts harvested from different autogenous areas or multiple non-autogenous materials as an alternative.

CAF combined with pSCTG is considered the gold standard for root coverage procedures. However, factors such as the density of vascular structures, a close approximation to nerves, and postoperative morbidity remain concerning for clinicians using palatal connective tissue grafts. Because of this, researchers have sought different techniques for palatal connective tissue harvesting and/or different autogenous donor areas. The maxillary tuberosity region has been found to have a denser lamina propria and is farther from nerve/vascular bundles.

Despite differences in harvesting techniques, literature has presented similar root coverage outcomes, lesser post-operative bleeding, and pain for SCTGs harvested from the maxillary tuberosity (tSCTG) compared to pSCTG groups. Decreased post-operative pain after tSCTG harvesting could be explained by higher amounts of connective tissue present in the donor area after harvesting and avoiding trauma created by food consumption and tongue movements in the region. Clinical data also showed an increased amount of keratinized tissue and its stability after augmentation, favoring tSCTG. Considering structural differences, literature has shown that tSCTG provides more thickness, a more abundant lamina propria, and denser collagen compared to pSCTG. However, due to the size of the harvested tSCTG not being as abundant as pSCTG, it can be assumed that the augmented areas were limited to multiple recessions or defects.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker, systemically healthy
* No active periodontal disease
* Maxillary anterior and premolar teeth with single, isolated recessions RT 1 (Miller 1 &2)
* Absences of non-carious cervical lesions (NCCL) and non-detectable cemento-enamel junction (CEJ)
* Buccal gingival recession defects between 2-5 mm in depth

Exclusion Criteria:

* Presence of caries lesions or restorations in the cervical area
* Intake of medications that impede periodontal tissue health and healing
* Medical contraindications for periodontal surgical procedures
* Pregnancy and lactation
* Bleeding and plaque scores ≥ 20%
* Probing depths > 4 mm

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of root coverage | 1-year postoperative follow-up
  Mean root coverage of tSCTG versus pSCTG with CAF according to the gingival recession changes from baseline and the 1-year postoperative follow-up

SECONDARY OUTCOMES:
The percentage of complete root coverage | 1-year postoperative follow-up
  After the 1-year postoperatively, absence of gingival recession
Recession depth | 1-year postoperative follow-up
  The distance between cemento-enamel junction and gingival margin
Patient morbidity - Postoperative pain | Up to 28 days postoperatively
  Postoperative pain will be assessed using a visual analogue score
Patient morbidity - Postoperative discomfort | Up to 28 days postoperatively
  Postoperative discomfort will be assessed using a visual analogue score
Histological features of the graft | Through study completion, an average of 1 year
  Graft cellularity
Histomorphometrical features of the graft | Through study completion, an average of 1 year
  The amount of lamina propria

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zucchelli G, Amore C, Sforza NM, Montebugnoli L, De Sanctis M. Bilaminar techniques for the treatment of recession-type defects. A comparative clinical study. J Clin Periodontol. 2003 Oct;30(10):862-70. doi: 10.1034/j.1600-051x.2003.00397.x. PMID 14710766
- [Background] Chambrone L, Tatakis DN. Periodontal soft tissue root coverage procedures: a systematic review from the AAP Regeneration Workshop. J Periodontol. 2015 Feb;86(2 Suppl):S8-51. doi: 10.1902/jop.2015.130674. PMID 25644302
- [Background] Jung UW, Um YJ, Choi SH. Histologic observation of soft tissue acquired from maxillary tuberosity area for root coverage. J Periodontol. 2008 May;79(5):934-40. doi: 10.1902/jop.2008.070445. PMID 18454674
- [Background] Zucchelli G, Mele M, Stefanini M, Mazzotti C, Marzadori M, Montebugnoli L, de Sanctis M. Patient morbidity and root coverage outcome after subepithelial connective tissue and de-epithelialized grafts: a comparative randomized-controlled clinical trial. J Clin Periodontol. 2010 Aug 1;37(8):728-38. doi: 10.1111/j.1600-051X.2010.01550.x. Epub 2010 Jun 24. PMID 20590963